CLINICAL TRIAL: NCT01229839
Title: Chemoembolization of Unresectable Hepatocellular Carcinoma With or Without Mixing the Chemotherapy With Lipiodol: Effectiveness and Safety. A Prospective and Randomized Clinical Trial.
Brief Title: Chemoembolization With or Without Mixing the Chemotherapy With Lipiodol for Unresectable HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: HCC_S010
Record Dates: First submitted 2010-10-25; First posted 2010-10-28 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma,Hepatocellular; Liver Neoplasms; Therapeutic; Chemoembolization,; TACE; pharmacokinetics; Iodized Oil/administration & dosage; polyvinyl alcohol; Humans
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Embolization, Therapeutic; Ethiodized Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- infusion group (Experimental): Infusion of anticancer agent followed by Embolization
  Interventions: Other: Embolization; Other: Infusion of anticancer agent
- lipiodol chemotherapy group (Experimental): Infusion of mixture of anticancer agent and lipiodol followed by Embolization
  Interventions: Other: Embolization; Other: Infusion of mixture of anticancer agent and lipiodol

INTERVENTIONS:
Other: Embolization — embolization with lipiodol and polyvinyl alcohol particles (PVA)
Other: Infusion of anticancer agent — infusion with chemotherapy drugs (EADM 50mg, lobaplatin 50mg, and MMC 6mg ) desolved in water
  Arms: infusion group
Other: Infusion of mixture of anticancer agent and lipiodol — infusion of mixture of lipiodol and chemotherapy drugs (EADM 50mg, lobaplatin 50mg, and MMC 6mg)dissolved in water-soluble contrast medium and distilled water
  Arms: lipiodol chemotherapy group

SUMMARY:
TACE is considered the standard treatment for unresectable HCC on the basis of the fact that there are no alternative to curative procedures.But the optimal combined regimen is still unclear. One of the controversy is do the protocol should contain lipiodo and how to executer. The investigators hypothesize that TACE without mixing the chemotherapy with lipiodol is not unacceptably worse than TACE mixing the chemotherapy with lipiodol.

ELIGIBILITY:
Eligibility criteria:

Inclusion Criteria:

* Adults patients with a diagnosis of HCC which is not amenable to surgical resection ,local ablative therapy and any other cured treatment.
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria. And the lesion has not been previously treated with TACE, surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* No serious concurrent medical illness
* Unresectable BCLC stage A-B disease
* No cirrhosis or cirrhotic status of Child-Pugh class A
* No significant renal impairment (creatinine clearance < 30 mL/minute) or patients on dialysis
* No current infections requiring antibiotic therapy
* Not on anticoagulation or suffering from a known bleeding disorder
* No unstable coronary artery disease or recent MI
* The following laboratory parameters:

  * Platelet count ≥ 60,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 1.5 mg/dL Serum albumin ≥ 35 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Known history of HIV
* History of organ allograft
* Pregnant or breast-feeding patients
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* severe Arterioportal Shunts or Arteriavein Shunts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 year

SECONDARY OUTCOMES:
Time to progression | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Caturelli E, Siena DA, Fusilli S, Villani MR, Schiavone G, Nardella M, Balzano S, Florio F. Transcatheter arterial chemoembolization for hepatocellular carcinoma in patients with cirrhosis: evaluation of damage to nontumorous liver tissue-long-term prospective study. Radiology. 2000 Apr;215(1):123-8. doi: 10.1148/radiology.215.1.r00ap21123. PMID 10751477
- [Background] Higashi S, Tabata N, Kondo KH, Maeda Y, Shimizu M, Nakashima T, Setoguchi T. Size of lipid microdroplets effects results of hepatic arterial chemotherapy with an anticancer agent in water-in-oil-in-water emulsion to hepatocellular carcinoma. J Pharmacol Exp Ther. 1999 May;289(2):816-9. PMID 10215657
- [Background] Madden MV, Krige JE, Bailey S, Beningfield SJ, Geddes C, Werner ID, Terblanche J. Randomised trial of targeted chemotherapy with lipiodol and 5-epidoxorubicin compared with symptomatic treatment for hepatoma. Gut. 1993 Nov;34(11):1598-600. doi: 10.1136/gut.34.11.1598. PMID 8244149
- [Background] Bruix J, Llovet JM, Castells A, Montana X, Bru C, Ayuso MC, Vilana R, Rodes J. Transarterial embolization versus symptomatic treatment in patients with advanced hepatocellular carcinoma: results of a randomized, controlled trial in a single institution. Hepatology. 1998 Jun;27(6):1578-83. doi: 10.1002/hep.510270617. PMID 9620330
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Ono Y, Yoshimasu T, Ashikaga R, Inoue M, Shindou H, Fuji K, Araki Y, Nishimura Y. Long-term results of lipiodol-transcatheter arterial embolization with cisplatin or doxorubicin for unresectable hepatocellular carcinoma. Am J Clin Oncol. 2000 Dec;23(6):564-8. doi: 10.1097/00000421-200012000-00006. PMID 11202797